CLINICAL TRIAL: NCT04538040
Title: An Open Label Study Evaluating the Safety and Efficacy of Switching From Rilpivirine/Emtricitabine/Tenofovir Alafenamide in Combination With Dolutegravir, to Bictegravir/Emtricitabine/Tenofovir Alafenamide in Combination With Doravirine, in Male HIV+ Subjects > 45 Years With Multi-drug Resistant Virus and Virologic Suppression (Documented With at Least One Viral Load Result < 50 Copies Per mL) During the Last 6 Months on Current Therapy
Brief Title: Bictegravir/Emtricitabine/Tenofovir Alafenide Plus Doravirine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Quest Clinical Research (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BETD-001
Record Dates: First submitted 2020-08-26; First posted 2020-09-03 (Actual); Results first posted 2024-03-05 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: HIV-1-infection
Keywords: multi-drug resistant
MeSH Terms: interventions — bictegravir; emtricitabine tenofovir alafenamide; bictegravir, emtricitabine, tenofovir alafenamide, drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Biktarvy + Doravirine Switch (Experimental): bictegravir 50mg/emtricitabine 200mg/tenofovir alafenamide 25mg tablets + doravirine 100mg tablets taken orally once per day
  Interventions: Drug: Bictegravir/emtricitabine/tenofovir alafenamide + Doravirine switch

INTERVENTIONS:
Drug: Bictegravir/emtricitabine/tenofovir alafenamide + Doravirine switch — Safety and efficacy of switching from rilpivirine/emtricitabine/tenofovir alafenamide in combination with dolutegravir, to bictegravir/emtricitabine/tenofovir alafenamide in combination with doravirine in male, 45+ year old subjects. The study will also include secondary outcomes of quality of life (QOL) and weight changes.
  Other Names: Biktarvy + Pifeltro Switch

SUMMARY:
The current study proposal is an open label observational trial for maintenance of virologic suppression, and is designed as a non- inferiority switch trial. The study will involve approximately 30 patients, which includes a PK arm of approximately 10 patients. The study will also include secondary outcomes of quality of life (QOL) and weight changes

Hypothesis:

Patients with prior NUC or NNRTI resistance (but not to rilpivirine or doravirine) will maintain their virologic suppression after a drug regimen switch from rilpivirine/emtricitabine/tenofovir alafenamide in combination with dolutegravir, to bictegravir/emtricitabine/tenofovir alafenamide in combination with doravirine. The switch therapy will avoid food interactions, and will be well tolerated by subjects.

ELIGIBILITY:
Inclusion Criteria:

* HIV positive Males, age 45 or older
* Any genotypic or phenotypic resistance except k65R, 69 insertion, integrase resistance, or resistance to rilpivarine or doravirine.
* Receiving combination antiretroviral regimen of rilpivirine/emtricitabine/tenofovir alafenamide in combination with dolutegravir > 12 months and with viral load <50 copies/ mL on at least one occasion within the six months prior to switch.
* Suppressed viral load as defined by one plasma HIV RNA level < 50 copies/mL within previous 6 months.
* Capable of providing informed consent

Exclusion Criteria:

* Any current or prior integrase inhibitor resistance
* Nucleoside reverse transcriptase (NRTI) mutation 69 insertion or k65R mutation
* Documented second generation non-nucleoside reverse transcriptase inhibitor (NNRTI) resistance (rilpivirine or doravirine)

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-12-19 (Actual); Primary Completion 2021-11-11 (Actual); Study Completion 2021-11-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- SFOMG Private Practice, San Francisco, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Biktarvy + Doravirine Switch
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Biktarvy + Doravirine Switch
Number analyzed (Participants) | 20
Age, Continuous [Median (Full Range); unit: years] | 65 [46 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 19
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Viral Suppression
Description: Percentage of patients with viral HIV load (VL) <50 and <200 copies/mL at 48 weeks
Time Frame: 48 Weeks
Measure: Number; unit: percentage of participants
Arm/Group | Biktarvy + Doravirine Switch
Number analyzed (Participants) | 20
percentage of participants | 100

2. Secondary Outcome: Tolerability of Study Drug
Description: Tolerability of study drugs will be assessed by summarizing the number of AE/SAEs occurring during the study
Time Frame: Week 48
Measure: Number; unit: Adverse Events
Arm/Group | Biktarvy + Doravirine Switch
Number analyzed (Participants) | 20
Adverse Events | 16

3. Secondary Outcome: Change in Body Mass Index
Description: Assess changes in BMI due to treatment switch
Time Frame: Week 48
Measure: Mean (Standard Deviation); unit: kg/m2
Arm/Group | Biktarvy + Doravirine Switch
Number analyzed (Participants) | 20
kg/m2 | -0.2 (.85)

4. Secondary Outcome: Work Productivity and Activity
Description: Improvement in work productivity and activity as measured by Work Productivity and Activity Impairment Questionnaire (WPAI). The range of the scale is 0-10, where 0 means it did not have an affect and 10 means it did have an affect.
Time Frame: Week 48
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Biktarvy + Doravirine Switch
Number analyzed (Participants) | 20
score on a scale
  Hours of Work Missed | 0 [0 to 10]
  Health Problem Affecting Productivity | 0 [0 to 5]
  Health Problems Affect on Daily Activities | 0 [0 to 10]

5. Secondary Outcome: PK Assessment
Description: Subject plasma concentration-time data of bictegravir and doravirine will be analyzed using non-compartmental model (WinNonlin®)
Time Frame: Week 4 (+/- 14 days) with time points at predose (-0.5 hr), 0.5, 1, 2, 4, 6, 8, 12, and 24 hours
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/ml
Arm/Group | Biktarvy + Doravirine Switch
Number analyzed (Participants) | 20
ug/ml
  Plasma BIC Cmax | 8.55 (33)
  Plasma DOR Cmax | 1.2 (34)

6. Secondary Outcome: Adverse Events Assessment
Description: Assess AE's of any grade and relationship to the drug combination occurring in at least 5% of participants or more.
Time Frame: Day 28, Weeks 12, 24, 36, & 48
Measure: Number; unit: Number of AEs
Arm/Group | Biktarvy + Doravirine Switch
Number analyzed (Participants) | 20
Number of AEs
  Mild Adverse Events | 14
  Moderate Adverse Events | 1
  Severe Adverse Events | 1

7. Secondary Outcome: Wellbeing Improvement
Description: Improvement in well-being and sleep inventory as measured by The Pittsburgh Sleep Quality Index (PSQI). Minimum score is 0 and maximum score is 21. A higher score indicates worse quality sleep.
Time Frame: Week 48
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Biktarvy + Doravirine Switch
Number analyzed (Participants) | 20
score on a scale | 7 [1 to 15]

ADVERSE EVENTS:
Time Frame: AE data is collected from the screening visit, and up to 30 days after the last dose of study drug, up to 48 weeks.
Arm/Group | Biktarvy + Doravirine Switch
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 11/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Biktarvy + Doravirine Switch (N=20)
New Onset Diabetes Mellitus (Metabolism and nutrition disorders) | 1 (1)
Intermittent Headache (General disorders) | 2 (2)
Renal Cell Carcinoma Removal (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Episode of Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Urinary Tract Infection (Renal and urinary disorders) | 1 (2)
Viral Load of 330 (Blood and lymphatic system disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Loose Stool (Gastrointestinal disorders) | 1 (1)
Arthritis in Right Hand (Musculoskeletal and connective tissue disorders) | 1 (1)
Abdominal Pain (General disorders) | 1 (1)
Hypertension (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Neck Sprain (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-06-25): https://cdn.clinicaltrials.gov/large-docs/40/NCT04538040/Prot_SAP_002.pdf
  • Informed Consent Form (2021-07-13): https://cdn.clinicaltrials.gov/large-docs/40/NCT04538040/ICF_001.pdf